CLINICAL TRIAL: NCT02560844
Title: Cardiomyopathy Arrhythmia Risk Evaluation
Acronym: CARE
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 08-0638
Record Dates: First submitted 2015-09-21; First posted 2015-09-25 (Estimated); Last update posted 2019-10-02 (Actual); Status verified 2017-10

CONDITIONS: Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will evaluate the prognostic utility of novel ECG markers of electrical instability in patients with cardiomyopathy.

DETAILED DESCRIPTION:
Baseline ECG markers of electrical instability will be measured in patients with cardiomyopathy. These ECG markers will be evaluated from a clinical Holter recording. All patients will have a primary implantable cardioverter defibrillator (ICD) as part of their clinical care. Patients will be followed prospectively for 2 years to evaluate the primary outcome of appropriate ICD shocks. Multivariable modelling will be performed to determine whether the ECG markers of electrical instability independently predict the primary clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* cardiomyopathy, primary prevention ICD

Exclusion Criteria:

* brady-pacing requirement

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cardiomyopathy and primary prevention ICDs
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2015-07; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with appropriate implantable cardioverter defibrillator (ICD) shocks | 2 years
  Proportion is from 0 (no patients with shocks) to 100% (all patients receive shocks)

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Suszko AM, Chakraborty P, Viswanathan K, Barichello S, Sapp J, Talajic M, Laksman Z, Yee R, Woo A, Spears D, Adler A, Rakowski H, Chauhan VS. Automated Quantification of Abnormal QRS Peaks From High-Resolution ECGs Predicts Late Ventricular Arrhythmias in Hypertrophic Cardiomyopathy: A 5-Year Prospective Multicenter Study. J Am Heart Assoc. 2022 Dec 6;11(23):e026025. doi: 10.1161/JAHA.122.026025. Epub 2022 Nov 29. PMID 36444865
- [Derived] Chakraborty P, Suszko AM, Viswanathan K, Sheikholeslami K, Spears D, Adler A, Woo A, Rakowski H, Chauhan VS. Microvolt QRS Alternans in Hypertrophic Cardiomyopathy: A Novel Risk Marker of Late Ventricular Arrhythmias. J Am Heart Assoc. 2021 Dec 7;10(23):e022036. doi: 10.1161/JAHA.121.022036. Epub 2021 Dec 2. PMID 34854315